CLINICAL TRIAL: NCT00690313
Title: To Compare the Efficacy of Topical Vigamox Eye Drops at Tid 3 Days Prior to Intravitreal Injection Versus Tid 1 Day Prior to Intravitreal Injection
Brief Title: Dosage Study for Vigamox Eye Drops Prior to Intravitreal Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Illinois Retina Associates (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vig508
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Intravitreal Injection Patients
Keywords: Vigamox, topical antibiotics, Intravitreal injections, macular degeneration, endophthalmitis
MeSH Terms: conditions — Macular Degeneration; Endophthalmitis | interventions — Moxifloxacin

ARMS (2):
- Arm 1 (Active Comparator): Arm 1: receives Vigamox eye drops 3Xday for 3 days prior to intravitreal injection
  Interventions: Drug: Vigamox
- Arm 2 (Active Comparator): Arm 2: receives Vigamox eye drops 3Xday for 1 day prior to intravitreal injection
  Interventions: Drug: Vigamox

INTERVENTIONS:
Drug: Vigamox — eye drops 3 times day either 1 or 3 days prior to intravitreal injection

SUMMARY:
Antibiotic eye drops are being used before and after intravitreal injections. Currently there is no study indicating the benefit of there usage or their dosage.

In this study we compare the efficacy of Vigamox eye drops (antibiotic)starting 3 days prior to the injection versus 1 day prior to intravitreal injection.

ELIGIBILITY:
Inclusion Criteria:

* Patient who need intravitreal injections patients who are willing to participate in the study

Exclusion Criteria:

* Patients who are allergic to Vigamox or who have taken any eye drops within the past 3 weeks

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Timed study | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kourous A Rezaei, MD, Principal Investigator — Illinois Retina Associates SC
Locations (1):
- Illinois Retina Associates, Harvey, Illinois, United States